CLINICAL TRIAL: NCT02916212
Title: Quality Improvement - Monitoring Alarm Optimization Study
Acronym: QI-MAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00073369
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2016-09

CONDITIONS: No Applicable Condition; Study of Physiologic Monitor Alarms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Hospital units where alarms have been optimized
  Interventions: Other: Optimized alarm profiles
- Control (No Intervention): Hospital units where alarms remain unchanged

INTERVENTIONS:
Other: Optimized alarm profiles
  Arms: Experimental

SUMMARY:
This project aims to reduce the frequency of duplicate, false and clinically insignificant alarms in hospital units, and subsequent alarm fatigue resulting from excessive alarm frequency. The investigators will implement evidence-based guidelines for alarm optimization according to patient-population specific parameters, and evaluate alarm frequency and staff perception of alarm fatigue at baseline and 60 days after implementation of this quality improvement initiative.

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff at selected units at Duke University Hospital

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of frequency of total alarms by hospital unit at 60 days | At baseline and 60 days following implementation

SECONDARY OUTCOMES:
Change from baseline of number of alarms per bed | At baseline and 60 days following implementation
Change from baseline of number of alarms per day per bed | At baseline and 60 days following implementation
Change from baseline of perceived alarm fatigue, assessed using a questionnaire | At baseline and 60 days following implementation